CLINICAL TRIAL: NCT06054893
Title: An Open-Label, Phase 1, Study to Evaluate the Pharmacokinetics, Safety, Tolerability, Pharmacodynamics, and Efficacy of Omaveloxolone in Participants ≥2 to <16 Years of Age With Friedreich's Ataxia
Brief Title: A Study to Find Out How BIIB141 (Omaveloxolone) is Processed in the Body and to Learn More About Its Safety in Participants With Friedreich's Ataxia Aged 2 to 15 Years Old
Acronym: BOLD
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 408-C-2001
Record Dates: First submitted 2023-09-13; First posted 2023-09-26 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Friedreich Ataxia
Keywords: Friedreich's ataxia; FA; RTA 408; Omaveloxolone
MeSH Terms: conditions — Friedreich Ataxia | interventions — omaveloxolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part 1 and 2: Cohort A1 (Experimental): Cohort A1 will contain participants 12 to <16 years of age. Participants will receive a single oral dose of omaveloxolone, 150 milligrams (mg), capsule, on Day 1 of the treatment period of part 1, followed by the same dose in part 2 up to week 240 or commercial availability whichever comes first. The dose in part 2 may be adjusted as per additional safety and Bayesian population pharmacokinetics (popPK) analyses.
  Interventions: Drug: Omaveloxolone
- Part 1 and 2: Cohort A2 (Experimental): Cohort A2 will contain participants 12 to <16 years of age. Participants will receive a single oral dose of omaveloxolone, capsule, at a dosage level determined by a Bayesian popPK analysis using the data from Cohort A1 to select the dose in part 1, followed by the same dose in part 2 up to week 240 or commercial availability whichever comes first. The dose in part 2 may be adjusted as per additional safety and Bayesian popPK analyses.
  Interventions: Drug: Omaveloxolone
- Part 1 and 2: Cohort B1 (Experimental): Cohort B1 will contain participants 7 to <12 years of age and will initiate in parallel with Cohort A2. Participants will receive a single oral dose of omaveloxolone, capsule, at a dosage level determined by a Bayesian popPK analysis using the data from Cohort A1 to select the dose in part 1, followed by the same dose in part 2 up to week 240 or commercial availability whichever comes first. The dose in part 2 may be adjusted as per additional safety and Bayesian popPK analyses.
  Interventions: Drug: Omaveloxolone
- Part 1 and 2: Cohort C1 (Experimental): Cohort C1 will contain participants 2 to <7 years of age. Participants will receive a single oral dose of omaveloxolone, capsule, at a dosage level determined by a Bayesian popPK analysis using the data from cohorts A1, A2, and B1 to select the dose in part 1, followed by the same dose in part 2 up to week 240 or commercial availability whichever comes first. The dose in part 2 may be adjusted as per additional safety and Bayesian popPK analyses.
  Interventions: Drug: Omaveloxolone
- Part 1 and 2: Cohort A3 (Experimental): Cohort A3 will contain participants 12 to <16 years of age. Participants will receive a single oral dose of omaveloxolone, capsule, at a dosage level determined by a Bayesian popPK analysis using the data from cohorts A1, A2, and B1 to select the dose in part 1, followed by the same dose in part 2 up to week 240 or commercial availability whichever comes first. The dose in part 2 may be adjusted as per additional safety and Bayesian popPK analyses.
  Interventions: Drug: Omaveloxolone
- Part 1 and 2: Cohort B2 (Experimental): Cohort B2 will contain participants 7 to <12 years of age and will initiate in parallel with Cohort A3. Participants will receive a single oral dose of omaveloxolone, capsule, at a dosage level determined by a Bayesian popPK analysis using the data from cohorts A1, A2, and B1 to select the dose in part 1, followed by the same dose in part 2 up to week 240 or commercial availability whichever comes first. The dose in part 2 may be adjusted as per additional safety and Bayesian popPK analyses.
  Interventions: Drug: Omaveloxolone
- Part 1 and 2: Cohort C2 (Experimental): Cohort C2 will contain participants 2 to <7 years of age. Participants will receive a single oral dose of omaveloxolone, capsule, at a dosage level determined by a Bayesian popPK analysis using the data from Cohorts A1, A2, A3, B1, B2, and C1 to select the dose in part 1, followed by the same dose in part 2 up to week 240 or commercial availability whichever comes first. The dose in part 2 may be adjusted as per additional safety and Bayesian popPK analyses.
  Interventions: Drug: Omaveloxolone

INTERVENTIONS:
Drug: Omaveloxolone — Administered as specified in the treatment arm
  Other Names: RTA 408; SKYCLARYS; BIIB141

SUMMARY:
In this study, researchers will learn more about BIIB141, also known as omaveloxolone or SKYCLARYS®. This drug has been approved, or made available for doctors to prescribe, for people with Friedrich's Ataxia (FA) who are at least 16 years old. But, it is not yet available for children and teens with FA who are younger than 16 years old. The main objective of this study is to learn how BIIB141 is processed in the body of children and teens who are 2 to 15 years old.

The main question researchers want to answer in this study is:

* How does the body process BIIB141 in children and teens?
* How many participants have medical problems during the study?
* Are there any changes in the participants' overall health during the study?
* Are there any changes in the participants' heart health?
* Are there any changes in how the participants move through puberty? Puberty is the time in someone's life when their body changes from a child to an adult.

This study will be done as follows:

* Participants will be screened to see if they can join the study. The screening period will be up to 14 days, after which participants will check into their study research center.
* There are 2 parts to this study. During Part 1, participants will take a single dose of BIIB141. Participants will be in 1 of 7 different groups based on their age:
* Group A1: 12 to 15 years old, taking 150 milligrams (mg) of BIIB141
* Group A2: 12 to 15 years old, taking a dose of BIIB141 based on the data from Group A1
* Group B1: 7 to 11 years old, taking a dose of BIIB141 based on Group A1 data
* Group C1: 2 to 6 years old, taking a dose of BIIB141 based on Groups A1, A2, and B1 data
* Group A3: 12 to 15 years old, taking a dose of BIIB141 based on Groups A1, A2, and B1 data
* Group B2: 7 to 11 years old, taking a dose of BIIB141 based on Groups A1, A2, and B1 data
* Group C2: 2 to 6 years old, taking a dose of BIIB141 based on Group A1, A2, A3, B1, B2, and C1 data.
* During Part 2, participants from Part 1 will take BIIB141 once in the study research center. Cohort A1 will take 150 mg of BIIB141. Dose of Cohorts A2 and B1 will be based on data from Cohort A1, dose of Cohorts C1, A3 and B2 will be based on data from Cohorts A1, A2 and B1, while Cohort C2's dose will be based on all the other groups. Participants will then take it once a day at home.
* After leaving the study research center in Part 2, participants will return for tests at Week 4, Week 12, Week 24, and then every 24 weeks. Participants will also be contacted by telephone at Week 2, Week 8, and Week 18.
* Participants will be in this study for up to 240 weeks.

DETAILED DESCRIPTION:
Recruitment will be limited to the U.S. only as participants will be able to remain on Part 2 of the study until they turn 16 and can access commercially-available drug which is FDA approved for age 16 and above. The part 1 primary objective of the study is to evaluate the pharmacokinetics (PK) of omaveloxolone following administration of a single dose in 3 age cohorts (2 to <7 years, 7 to <12 years, and 12 to <16 years) and secondary objective is to evaluate safety and tolerability of drug. The part 2 primary objective is to evaluate long term safety and tolerability of omaveloxolone.

ELIGIBILITY:
Part 1:

Inclusion Criteria:

* Have genetically confirmed FA.
* Have a left ventricular ejection fraction ≥ 40% (based on ECHO performed at Screening Visit).
* During screening, during the treatment period, and until 28 days following administration of the last dose of omaveloxolone, females of childbearing potential must practice at least 1 of the acceptable methods of birth control.
* During screening, during the treatment period, and until 28 days after the last dose of omaveloxolone, fertile males who have female partners of childbearing potential must practice one of the acceptable methods of birth control.

Exclusion Criteria:

* Have uncontrolled diabetes (haemoglobin A1c [HbA1c] >11.0%).
* Have B-type natriuretic peptide (BNP) level >200 picograms per milliliter (pg/mL) at screening.
* Have a history of clinically significant (CS) left-sided heart disease and/or CS cardiac disease, with the exception of mild to moderate cardiomyopathy associated with FA.
* Presence of outflow tract obstruction defined as a peak instantaneous gradient >50 mmHg (based on ECHO performed at screening).
* Have taken any moderate or strong inhibitors and/or inducers of cytochrome P450 3A4 within the 7 days prior to Day 1 or plan to take during study participation (eg, itraconazole, carbamazepine, phenytoin, ciprofloxacin, grapefruit juice, cannabidiol, fluconazole, fluvoxamine, verapamil, diltiazem).
* Have a history of CS liver disease (eg, fibrosis, cirrhosis, hepatitis), or have clinically relevant deviations in laboratory tests at screening
* Plan to or have participated in any other interventional clinical study within the 30 days prior to Day 1.
* Have a cognitive impairment that may preclude ability to comply with study procedures, in the opinion of the investigator.
* Be unable to comply with the requirements of the study protocol or be unsuitable for the study for any reason, in the opinion of the investigator.
* Have previously documented mitochondrial respiratory chain disease.
* Have a history of thromboembolic events within the past 5 years.
* Plan to or have taken anticoagulant therapy within 30 days prior to Day 1 with the exception of a daily low dose aspirin (up to 81 mg).
* Plan to or have scheduled surgical treatment for scoliosis or foot deformity during the study.
* Have had significant suicidal ideation within 30 days prior to Screening Visit, as per investigator judgment, or any history of suicide attempt.
* For females, be pregnant or breastfeeding.

Part 2:

* No discontinuation criteria have been met.
* Safety and tolerability data from Part 1 are supportive of continuation in the judgement of the Investigator.

In the event of intercurrent illness or other change in health status of the participant, additional Part 1 Screening assessments may be repeated prior to initiation of Part 2, based on the judgement of the Investigator in consultation with the Medical Monitor.

NOTE: Other protocol- defined Inclusion/Exclusion criteria may apply.

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2030-02-21 (Estimated); Study Completion 2030-11-22 (Estimated)

PRIMARY OUTCOMES:
Part 1: Apparent Clearance (CL/F) of Omaveloxolone | Predose (0 hour), after dose 1 hour, 2 hours, 3 hours, 4 hours, 24 hours, and 96 hours
Part 1: Maximum Concentration (Cmax) of Omaveloxolone | Predose (0 hour), after dose 1 hour, 2 hours, 3 hours, 4 hours, 24 hours, and 96 hours
Part 1: Volume of Distribution (V/F) of Omaveloxolone | Predose (0 hour), after dose 1 hour, 2 hours, 3 hours, 4 hours, 24 hours, and 96 hours
Part 1: Area Under the Plasma Concentration-Time Curve From 0 Extrapolated to Infinity (AUC0-∞) of Omaveloxolone | Predose (0 hour), after dose 1 hour, 2 hours, 3 hours, 4 hours, 24 hours, and 96 hours
Part 1: Area Under the Plasma Concentration-Time Curve From 0 to tlast (AUC0-tlast) of Omaveloxolone | Predose (0 hour), after dose 1 hour, 2 hours, 3 hours, 4 hours, 24 hours, and 96 hours
Part 1: Area Under the Plasma Concentration-Time Curve From 0 to 24 Hours (AUC0-24) of Omaveloxolone | Predose (0 hour), after dose 1 hour, 2 hours, 3 hours, 4 hours, 24 hours, and 96 hours
Part 1: Individual Steady-State AUC0-24 (AUC0-24,ss) of Omaveloxolone | Predose (0 hour), after dose 1 hour, 2 hours, 3 hours, 4 hours, 24 hours, and 96 hours
Part 1: Individual Steady-State Cmax (Cmax,ss) of Omaveloxolone | Predose (0 hour), after dose 1 hour, 2 hours, 3 hours, 4 hours, 24 hours, and 96 hours
Part 1: Concentration at the end of a 24-Hour Dosing Interval (Ctrough,ss) of Omaveloxolone | Predose (0 hour), after dose 1 hour, 2 hours, 3 hours, 4 hours, 24 hours, and 96 hours
Part 2: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Day 1 up to the end of study (up to Week 240)
  An AE is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including abnormal laboratory finding), symptom, or disease temporally associated with use of a medicinal (investigational) product, whether or not related to medicinal (investigational) product. SAE is any untoward medical occurrence that at any dose results in death, in the view of investigator, places the participant at immediate risk of death (life-threatening event), requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, results in congenital anomaly/birth defect or is medically important event.
Part 2: Number of Participants With Clinically Significant Abnormality in Clinical Laboratory Assessments | From Day 1 up to Week 240
Part 2: Number of Participants With Clinically Significant Abnormality in Vital Signs | From Day 1 up to Week 240
  Vital signs, including blood pressure (BP), heart rate (HR), and oral body temperature, will be assessed.
Part 2: Number of Participants With Clinically Significant Abnormality in Electrocardiograms (ECGs) | From Day 1 up to Week 240
Part 2: Number of Participants With Change from Baseline in Echocardiogram (ECHO) | From Day 1 up to Week 240
Part 2: Number of Participants With Change from Baseline in Height | From Day 1 up to Week 240
Part 2: Number of Participants With Change from Baseline in Weight | From Day 1 up to Week 240
Part 2: Number of Participants With Change from Baseline Body Mass Index (BMI) | From Day 1 up to Week 240
Part 2: Number of Participants With Change from Baseline in Tanner Assessment | From Day 1 up to Week 240
Part 2: Number of Participants With Change from Baseline in Paediatric Growth (Height) | From Day 1 up to Week 240
Part 2: Number of Participants With Change from Baseline in Paediatric Growth (Weight) | From Day 1 up to Week 240

SECONDARY OUTCOMES:
Part 1: Number of Participants With AEs and SAEs | From Day 1 up to Day 22
Part 1: Number of Participants With Abnormality in Clinical Laboratory Assessments | From Day 1 up to Day 22
Part 1: Number of Participants With Abnormality in Vital Signs | From Day 1 up to Day 22
Part 1: Number of Participants With Abnormality in ECGs | From Day 1 up to Day 22

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/